CLINICAL TRIAL: NCT06787495
Title: Predictors of Limb Loss in Peripheral Arterial Trauma Patients
Brief Title: Limb Salvage in Peripheral Arterial Trauma Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Mekhael Rezk Abd-Elmalak (Other)
Responsible Party: Sponsor-Investigator, Mekhael Rezk Abd-Elmalak, Mekhael Rezk Abd-Elmalak Mesael, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Arterial trauma patients
Record Dates: First submitted 2025-01-11; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Trauma Patients
Keywords: Trauma patients with peripheral arterial trauma patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Arterial repair — Arterial repair starting from simple repair or vein graft or synthetic graft

SUMMARY:
The aim of this study is to determine risk factors associated with failure of limb salvage in patients with periphral arterial injuries with or without attempts of revascularization.

DETAILED DESCRIPTION:
Trauma to the vascular system can be devastating. Peripheral arterial traumatic injuries rarely occur in isolation, often complicated by bone fractures and nerve injuries. As a result of these complex injury patterns, vascular extremity trauma presents unique challenges to injury management and is associated with significant morbidity.

In all trauma- related injuries , trauma is now the third leading cause of death and number one cause of death in people between the ages of 1 and 44 years . Vascular injuries comprise 3% of all civilian trauma and have significant potential morbidity. Leg trauma is common. However, it is associated with a significant vascular injury.The high energy of crushing trauma can cause extensive tissue damage with detrimental outcome such as high morbidity and mortality.[3] Management of associated life-threatening injuries takes priority which might lead to delay in definitive vascular repairs with subsequent limb loss.The most important risk factor for early limb loss is failed revascularization which is time dependent

ELIGIBILITY:
Inclusion Criteria:

* peripheral arterial trauma patients

Exclusion Criteria:

* trauma patients with vascular injuries other than peripheral arteries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be : technical success of the surgical intervention to control the bleeding and maintain vascularity of the affected limb (2) predictors of limb salvage. | From January 2021 to December 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McAndrew MP, Lantz BA. Initial care of massively traumatized lower extremities. Clin Orthop Relat Res. 1989 Jun;(243):20-9. PMID 2721064
- [Background] Bondurant FJ, Cotler HB, Buckle R, Miller-Crotchett P, Browner BD. The medical and economic impact of severely injured lower extremities. J Trauma. 1988 Aug;28(8):1270-3. doi: 10.1097/00005373-198808000-00023. PMID 3137367
- [Background] Mullenix PS, Steele SR, Andersen CA, Starnes BW, Salim A, Martin MJ. Limb salvage and outcomes among patients with traumatic popliteal vascular injury: an analysis of the National Trauma Data Bank. J Vasc Surg. 2006 Jul;44(1):94-100. doi: 10.1016/j.jvs.2006.02.052. PMID 16828431
- [Background] Howe HR Jr, Poole GV Jr, Hansen KJ, Clark T, Plonk GW, Koman LA, Pennell TC. Salvage of lower extremities following combined orthopedic and vascular trauma. A predictive salvage index. Am Surg. 1987 Apr;53(4):205-8. PMID 3579025